CLINICAL TRIAL: NCT04254471
Title: Multicenter, Phase II/III Study of Carboplatin Plus Etoposide With AL3810 in Participants With Untreated Extensive-Stage (ES) Small Cell Lung Cancer (SCLC)
Brief Title: This Phase II/III, Multicenter Study is Designed to Evaluate the Safety and Clinical Activity of AL3810 in Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AL3810-301
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Rabeprazole; E-3810; EC regimen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation (AL3810 + carboplatin + etoposide) (Experimental): Phase II:Participants will receive AL3810 orally in combination with carboplatin and etoposide during the Cycles 1-4 . AL3810 dose escalated form 5mg to 10mg step-up to determine the recommended dose of AL3810 in combination with carboplatin plus (+) etoposide in untreated participants with ES-SCLC.
  Interventions: Drug: AL3810; Drug: carboplatin + etoposide
- AL3810+ carboplatin + etoposide (Experimental): Phase III:Participants will receive AL3810(recommended dose will be determined by safety monitoring committee (SMC) in Phase II) orally in combination with carboplatin and etoposide during the Cycles 1-4. Thereafter, participants will receive maintenance AL3810 until persistent radiographic PD, intolerable toxicity or withdrawal of consent, investigator's consideration, lost follow up, death ,study termination by the sponsor.whichever occurs first.
  Interventions: Drug: AL3810; Drug: carboplatin + etoposide
- Placebo+ carboplatin + etoposide (Placebo Comparator): Phase III:Participants will receive placebo orally in combination with carboplatin and etoposide during the induction Cycles 1-4. Thereafter, participants will receive maintenance placebo until persistent radiographic PD, intolerable toxicity or withdrawal of consent, investigator's consideration, lost follow up, death ,study termination by the sponsor.whichever occurs first.
  Interventions: Drug: carboplatin + etoposide; Drug: Placebo

INTERVENTIONS:
Drug: AL3810 — 5mgQD, 7.5mgQD, 10mgQD
  Other Names: Lucitanib; E3810; E-3810
  Arms: AL3810+ carboplatin + etoposide; Dose escalation (AL3810 + carboplatin + etoposide)
Drug: carboplatin + etoposide — Carboplatin and etoposide are background treatment.
Drug: Placebo — Placebo
  Arms: Placebo+ carboplatin + etoposide

SUMMARY:
Phase II Study is to Evaluate the Safety and tolerability of AL3810 in combination with carboplatin plus (+) etoposide in untreated participants with ES-SCLC.

Phase III Study is to Evaluate the efficacy of AL3810 in combination with carboplatin plus (+) etoposide in untreated participants with ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Male or female, 18 ~75years of age
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed ES-SCLC
* No prior treatment for ES-SCLC
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function.
* Serum pregnancy test in screening period for women of childbearing potential should be negative.Except for women who have a history of sterilization or are postmenopausal.Men or woman subjects of reproductive age and their partners must agree to use effective contraception for at least 6 months from the date of signing the Informed Consent Form(ICF) until the last dose of the investigational therapy.

exclusion criteria: main exclusion criteria

* Histologically confirmed mixed small cell lung cancer.
* Symptoms related to central nervous system(CNS) metastasis, unstable CNS metastasis, or CNS diseases needed the increase of steroid dosage to control.
* Uncontrolled hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 313 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2022-05-22 (Estimated); Study Completion 2022-11-22 (Estimated)

PRIMARY OUTCOMES:
Phase II:adverse event(AE)/serious adverse event(SAE) | From the date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  AE/SAE to find the recommended dose of AL3810
Phase III:1.PFS | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 56 months
  1. Duration of Progression-Free Survival (PFS) as Assessed by the Independent Review Committee Using RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China